CLINICAL TRIAL: NCT02331940
Title: Tiotropium Respimat Soft Mist Inhaler Versus HandiHaler to Improve Sleeping Oxygen Saturation and Sleep Quality in COPD.
Brief Title: Tiotropium Respimat Versus HandiHaler on SaO2 and Sleep in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Crete (Other)
Responsible Party: Principal Investigator, Izolde Bouloukaki, Consultant, University of Crete
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COPDTIOT100
Record Dates: First submitted 2015-01-03; First posted 2015-01-06 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; sleeping oxygen saturation; sleep quality
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Initiation and Maintenance Disorders | interventions — Tiotropium Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Handihaler (Active Comparator): Tiotropium was delivered by the HandiHaler® device, a single-dose dry powder inhaler
  Interventions: Drug: tiotropium; Device: Handihaler
- Respimat (Active Comparator): Tiotropium was delivered via the Respimat® Soft Mist Inhaler,
  Interventions: Drug: tiotropium; Device: Respimat

INTERVENTIONS:
Drug: tiotropium — Comparison of the effect of tiotropium delivered by the Respimat Soft Mist Inhaler versus the HandiHaler on sleeping oxygen saturation and sleep quality in patients with COPD.
  Other Names: Spiriva
Device: Handihaler — Inhalation via the HandiHaler once daily
  Arms: Handihaler
Device: Respimat — Inhalation via the Respimat once daily
  Arms: Respimat

SUMMARY:
The aim of this study was to compare the tiotropium Respimat Soft Mist Inhaler and the HandiHaler in terms of their effects on sleeping oxygen saturation (SaO2) and sleep quality in patients with COPD.

DETAILED DESCRIPTION:
Patients with chronic obstructive pulmonary disease (COPD) have poor sleep quality as a result of various alterations in oxygenation parameters and sleep macro- and micro-architecture. We aimed to compare the tiotropium Respimat Soft Mist Inhaler and the HandiHaler in terms of their effects on sleeping oxygen saturation (SaO2) and sleep quality in patients with COPD. In a randomized, parallel-group trial involving 200 patients with mild to moderate COPD (resting arterial oxygen tension >60 mmHg while awake), we compared the effects of 6 months' treatment with the two devices on sleeping SaO2 and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged >=40 years old
* current or ex-smokers with a smoking history of at least 10 pack-years
* mild to moderate stable COPD (Global Initiative for Chronic Obstructive Lung Disease [GOLD] Stage I and II according to the 2010 GOLD guidelines (a post-bronchodilator forced expiratory volume in the first second (FEV1) ≥80% of predicted for stage I and 50% ≤ FEV1 < 80% of predicted for stage II, with a post-bronchodilator FEV1/forced vital capacity (FVC) ratio <0.70 at screening)
* waking arterial oxygen tension (PaO2) ≥60 mmHg

Exclusion Criteria:

* refusal to participate
* respiratory tract infection within 4 weeks prior to screening
* COPD exacerbations requiring treatment with antibiotics and/or oral corticosteroids and/or hospitalization within 6 weeks prior to screening
* concomitant pulmonary diseases other than COPD
* asthma
* evidence of sleep apnea on baseline sleep studies
* obesity hypoventilation syndrome
* respiratory failure
* congestive heart failure
* a history of life-threatening arrhythmias
* cardiomyopathy
* long-QT syndrome or QTc >450 ms at screening
* diabetes
* long-term oxygen therapy
* symptomatic prostatic hyperplasia
* bladder-neck obstruction
* moderate/severe renal impairment
* urinary retention
* narrow-angle glaucoma
* family or personal history of mental illness
* drug or alcohol abuse
* severe cognitive impairment
* concurrent oncological diseases
* history of narcolepsy or restless legs syndrome
* known history of alpha-1 antitrypsin deficiency
* participation in the active phase of a supervised pulmonary rehabilitation program
* hypersensitivity to any of the test ingredients
* history of adverse reactions to inhaled anticholinergics.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-03; Primary Completion 2013-12 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sophia E Schiza, MD, PhD, Study Chair — University of Crete

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Handihaler | Respimat
Started | 100 | 100
Completed | 93 | 95
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Handihaler | Respimat | Total
Number analyzed (Participants) | 93 | 95 | 188
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.7 (11.3) | 54.9 (11.8) | 54.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 25 | 55
  Male | 63 | 70 | 133
Region of Enrollment [Number; unit: participants]
  Greece | 93 | 95 | 188

OUTCOME MEASURES:

1. Primary Outcome: Sleeping Oxygen Saturation
Description: Mean sleeping oxygen saturation (%)
Time Frame: 6 months after treatment initiation
Measure: Mean (Standard Deviation); unit: percentage of Oxygen Saturation
Arm/Group | Handihaler | Respimat
Number analyzed (Participants) | 93 | 95
percentage of Oxygen Saturation | 94.4 (2.4) | 94.4 (2.2)
Statistical Analysis 1: Comparison: Handihaler vs Respimat; Test type: Superiority or Other; p = 0.88, t-test, 1 sided — p<0.05 was considered statistically significant

2. Primary Outcome: Sleep Quality
Description: Sleep quality, meaning the architecture of sleep (amount of the different sleep stages across the sleep episode),consists of sleep efficiency (%) (total sleep time - TST divided by the total time in bed and multiplied by 100), REM (%TST) (rapid eye movement sleep divided by TST and multiplied by 100) and NREM (%TST) (non-rapid eye movement sleep divided by TST and multiplied by 100).
  NORMAL RANGES Sleep efficiency: Normal is approximately 85 to 90% or higher. NREM (%TST): 75-80% REM (%TST) normally occupies about 20-25% of sleep time.
Time Frame: 6 months after treatment initiation
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Handihaler | Respimat
Number analyzed (Participants) | 93 | 95
percentage of time
  sleep efficiency (%) | 73.2 (11.8) | 79.1 (13.4)
  NREM (%TST) | 87.3 (4.9) | 85.3 (5.2)
  REM (%TST) | 12.7 (4.9) | 14.7 (5.2)

3. Secondary Outcome: Sleepiness
Description: Sleepiness - Epworth Sleepiness Scale (ESS) score (range 0-24, higher values indicate worse outcome, >10 indicates sleepiness, >16 excessive sleepiness)
Time Frame: 6 months after treatment initiation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Handihaler | Respimat
Number analyzed (Participants) | 93 | 95
units on a scale | 6.5 (5.9) | 6.1 (5.8)

4. Secondary Outcome: Hospitalization Rate
Description: Number of patients needed hospitalization
Time Frame: 6 months after treatment initiation
Measure: Number; unit: participants
Arm/Group | Handihaler | Respimat
Number analyzed (Participants) | 93 | 95
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Handihaler | Respimat
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/95
Other Adverse Events (participants affected / at risk) | 0/93 | 0/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No